CLINICAL TRIAL: NCT00732615
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Investigate the Use of NPSP558, a Recombinant Human Parathyroid Hormone (rhPTH[1-84]) for the Treatment of Adults With Hypoparathyroidism
Brief Title: Use of NPSP558 in the Treatment of Hypoparathyroidism
Acronym: REPLACE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL1-11-040; 2008-005063-34 (EudraCT Number)
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Results first posted 2015-03-06 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Hypoparathyroidism
Keywords: Hypoparathyroidism
MeSH Terms: conditions — Hypoparathyroidism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Sterile water for injection
  Interventions: Drug: Placebo
- 50, 75, 100 mcg NPSP558 (Experimental): Initial dose of 50mcg, to be titrated up to 75mcg and then 100mcg dependent upon response
  Interventions: Drug: NPSP558

INTERVENTIONS:
Drug: Placebo — Placebo for subcutaneous injection
  Arms: Placebo
Drug: NPSP558 — Parathyroid hormone 50, 75, or 100 mcg injectable subcutaneously daily
  Arms: 50, 75, 100 mcg NPSP558

SUMMARY:
Use of PTH (1-84) a recombinant hormone in escalating doses for the treatment of adults with hypoparathyroidism. The use of PTH should result in a decrease of calcium and vitamin D supplements.

DETAILED DESCRIPTION:
Patients with a history of hypoparathyroidism will be randomized to receive placebo or study drug for 24 weeks, which will be injected daily in either thigh. During that time they will be monitored for safety (specifically, calcium levels in the blood and urine). In addition, the patients' intake of Vitamin D and calcium will be measured.

ELIGIBILITY:
Inclusion Criteria

Patients who meet all of the following inclusion criteria can be enrolled and potentially randomized into this study:

* Adult males or females 18 to 85 years of age (prior to screening)
* History of hypoparathyroidism for ≥ 18 months
* Requirement for vitamin D metabolite/analog therapy with calcitriol ≥0.25 μg per day or alphacalcidol ≥0.50 μg per day prior to randomization. Requirement for supplemental oral calcium treatment ≥ 1000 mg per day over and above normal dietary calcium intake
* Serum thyroid function tests within normal laboratory limits at screening
* Serum magnesium levels within laboratory normal limits
* Serum 25-hydroxyvitamin D [25(OH)D] level ≤ 1.5-fold the laboratory upper limit of normal
* Creatinine clearance > 30 mL/min on two separate measurements OR creatinine clearance > 60 mL/min AND serum creatinine < 1.5 mg/dL
* With regard to female patients: women who are postmenopausal and women who are surgically sterilized can be enrolled. Women of childbearing potential must have a negative pregnancy test at Randomization and be willing to use two medically acceptable methods of contraception for the duration of the study.

Exclusion Criteria

Patients who have any of the following during the screening visit are not eligible for enrollment in this study:

* Known history of hypoparathyroidism resulting from an activating mutation in the CaSR gene or impaired responsiveness to PTH (pseudohypoparathyroidism)
* Any disease that might affect calcium metabolism or calcium-phosphate homeostasis other than hypoparathyroidism, such as active hyperthyroidism, Paget's disease, insulin dependent diabetes mellitus (IDDM) or poorly controlled Type II diabetes mellitus (HbA1C > 8%), severe and chronic cardiac, liver or renal disease, Cushing's syndrome, neuromuscular disease such as rheumatoid arthritis, myeloma, pancreatitis, malnutrition, rickets, recent prolonged immobility, active malignancy, primary or secondary hyperparathyroidism, a history of parathyroid carcinoma, hypopituitarism, acromegaly, or multiple endocrine neoplasia types I and II
* Patients with a history of thyroid cancer must be documented to be disease-free for a period of at least 5 years
* Patients dependent on regular parenteral calcium infusions (eg calcium gluconate) to maintain calcium homeostasis
* Patients that have undergone gastric resection or have active peptic ulcer disease requiring medical therapy
* Use of prohibited medications such as loop and thiazide diuretics, raloxifene hydrochloride, lithium, estrogens and progestins for hormone replacement therapy,methotrexate, or systemic corticosteroids within respective prohibited periods
* Previous treatment with PTH-like drugs, including PTH(1-84), PTH(1-34) or other N-terminal fragments or analogs of PTH or PTH-related protein within 6 months prior to screening
* Other drugs known to influence calcium and bone metabolism, such as calcitonin, fluoride tablets, or cinacalcet hydrochloride within the prohibited period
* Use of oral bisphosphonates within the previous 6 months or IV bisphosphonate preparations within the previous 12 months prior to screening
* Seizure disorder/epilepsy with a history of a seizure within the previous 6 months prior to screening
* Presence of open epiphyses
* Irradiation (radiotherapy) to the skeleton within 5 years
* Serum 25-hydroxyvitamin D levels greater than 1.5-fold the laboratory upper limit of normal
* Participation in any other investigational trial in which receipt of investigational drug or device occurred within 6 months prior to screening for this study
* Pregnant or lactating women
* History of diagnosed drug or alcohol dependence within the previous 3 years
* Clinical history of renal calculi within the past 12 months
* History of gout
* Disease processes that may adversely affect gastrointestinal absorption, including but not limited to short bowel syndrome, bowel resection, tropical sprue, celiac disease, ulcerative colitis, and Crohn's disease
* Chronic/severe cardiac disease including but not limited to cardiac insufficiency, arrhythmias, bradycardia (resting heart rate < 60 beats/minute), or hypotension (systolic and diastolic blood pressures < 100 and 60 mmHg, respectively)
* History of cerebrovascular accident (CVA).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2008-12-18 (Actual); Primary Completion 2011-09-28 (Actual); Study Completion 2011-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (31):
- United States (19):
  - Mayo Clinic-Scottsdale, Scottsdale, Arizona
  - Advance Medical Research LLC, Lakewood, California
  - Diabetes Associates, Orange, California
  - University of California-San Francisco VA Medical Center, San Francisco, California
  - Palm Springs Research Institute, Hialeah, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Michigan Bone and Mineral Clinic PC, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Columbia University Medical Center, New York, New York
  - University Physicians Group, Staten Island, New York
  - Physicians East, Greenville, North Carolina
  - University of Cincinnati Bone Health and Osteoporosis Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cetero Research DGD Research Inc., San Antonio, Texas
  - Hillcrest Family Health Center, Waco, Texas
  - The Vancouver Clinic, Vancouver, Washington
- Chetre Hospitalier Universitaire de Liege, Liège, Belgium
- Canada (3):
  - Heritage Medical Research Clinic, Calgary, Alberta
  - Capital District Health Authority, QEII Health Sciences Centre, Halifax, Nova Scotia
  - Oakville Bone Center, Oakville, Ontario
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Odense University Hospital, Odense
- Hôpital Européen Georges Pompidou, Paris, France
- Hungary (3):
  - Semmelweis University Medical School, Budapest
  - University of Pécs, School of Medicine, Pécs
  - University of Szeged, Szeged
- University Hospital of Careggi, Florence, Italy
- Royal Liverpool University Hospital, Liverpool, United Kingdom

REFERENCES:
- [Derived] Ayodele O, Rejnmark L, Mu F, Lax A, Berman R, Swallow E, Gosmanova EO. Five-Year Estimated Glomerular Filtration Rate in Adults with Chronic Hypoparathyroidism Treated with rhPTH(1-84): A Retrospective Cohort Study. Adv Ther. 2022 Nov;39(11):5013-5024. doi: 10.1007/s12325-022-02292-1. Epub 2022 Aug 26. PMID 36018496
- [Derived] Rejnmark L, Ayodele O, Lax A, Mu F, Swallow E, Gosmanova EO. The risk of chronic kidney disease development in adult patients with chronic hypoparathyroidism treated with rhPTH(1-84): A retrospective cohort study. Clin Endocrinol (Oxf). 2023 Apr;98(4):496-504. doi: 10.1111/cen.14813. Epub 2022 Aug 28. PMID 35974422
- [Derived] Ayodele O, Mu F, Berman R, Swallow E, Rejnmark L, Gosmanova EO, Kaul S. Lower Risk of Cardiovascular Events in Adult Patients with Chronic Hypoparathyroidism Treated with rhPTH(1-84): A Retrospective Cohort Study. Adv Ther. 2022 Aug;39(8):3845-3856. doi: 10.1007/s12325-022-02198-y. Epub 2022 Jun 11. PMID 35696069
- [Derived] Chen KS, Gosmanova EO, Curhan GC, Ketteler M, Rubin M, Swallow E, Zhao J, Wang J, Sherry N, Krasner A, Bilezikian JP. Five-year Estimated Glomerular Filtration Rate in Patients With Hypoparathyroidism Treated With and Without rhPTH(1-84). J Clin Endocrinol Metab. 2020 Oct 1;105(10):e3557-65. doi: 10.1210/clinem/dgaa490. PMID 32738041
- [Derived] Vokes TJ, Mannstadt M, Levine MA, Clarke BL, Lakatos P, Chen K, Piccolo R, Krasner A, Shoback DM, Bilezikian JP. Recombinant Human Parathyroid Hormone Effect on Health-Related Quality of Life in Adults With Chronic Hypoparathyroidism. J Clin Endocrinol Metab. 2018 Feb 1;103(2):722-731. doi: 10.1210/jc.2017-01471. PMID 29099947
- [Derived] Mannstadt M, Clarke BL, Vokes T, Brandi ML, Ranganath L, Fraser WD, Lakatos P, Bajnok L, Garceau R, Mosekilde L, Lagast H, Shoback D, Bilezikian JP. Efficacy and safety of recombinant human parathyroid hormone (1-84) in hypoparathyroidism (REPLACE): a double-blind, placebo-controlled, randomised, phase 3 study. Lancet Diabetes Endocrinol. 2013 Dec;1(4):275-83. doi: 10.1016/S2213-8587(13)70106-2. Epub 2013 Oct 7. PMID 24622413

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 124 Subjects were enrolled between 12/2008 and 9/2011 at 28 clinical sites in North America, Western Europe and Hungary.
Pre-assignment Details: Subjects underwent a screening and stabilization period (optimization) of up to 16 weeks prior to enrollment. Please note: Data for 10 subjects were excluded.
Groups:
- Placebo: Matching Placebo: Placebo for subcutaneous injection
- NPSP558: NPSP558: Recombinant Human Parathyroid hormone (rhPTH[1-84]) 50, 75, or 100 mcg subcutaneously daily
Period: Overall Study
Arm/Group | Placebo | NPSP558
Started | 40 | 84
Completed | 33 | 79
Not Completed | 7 | 5
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 0 | 2
Not completed — Physician Decision | 3 | 0
Not completed — Non-Compliance, Subject/Physician Dec. | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | NPSP558 | Total
Number analyzed (Participants) | 40 | 84 | 124
Age, Customized [Count of Participants; unit: Participants]
  < 45 years | 13 | 35 | 48
  45 to 64 years | 23 | 45 | 68
  > = 65 years | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 65 | 98
  Male | 7 | 19 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 40 | 82 | 122
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 1 | 1
  White | 39 | 80 | 119
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  North America | 21 | 43 | 64
  Europe | 12 | 25 | 37
  Hungary | 7 | 16 | 23

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects Who Met the Triple Efficacy Endpoint Criteria at Week 24.
Description: The triple efficacy endpoint criteria were defined as at least a 50% reduction from the baseline in oral calcium dose and at least a 50% reduction from the baseline in active vitamin D dose and an albumin-corrected total serum calcium concentration that was maintained or normalized compared to the baseline value (≥ 7.5 mg/dL) and did not exceed the upper limit of the laboratory normal range. The analysis of primary efficacy endpoint was based on investigator prescribed data.
Time Frame: Week 24 of dosing
Population: Intent to Treat (ITT) population, which includes all randomized subjects who received at least 1 dose of study drug and had at least 1 post-baseline efficacy assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | NPSP558
Number analyzed (Participants) | 40 | 84
percentage of participants | 2.5 [0.1 to 13.2] | 54.8 [43.5 to 65.7]
Statistical Analysis 1: Comparison: Placebo vs NPSP558; The null hypothesis is that the % of subjects meeting primary efficacy endpoint criteria are the same for both tmt arms. The sample size was determined based on the assumption that 40% and 10% of subjects for NPSP558 and pbo arms would meet the endpt criteria, respectively. Based on 2-tailed test, alpha of 0.05 and 2-to-1 randomization ratio, 84 (56 NPSP558, 28 pbo) subjects who completing the study would achieve 80% statistical power. Adjusted for dropouts, planned enrollment was 110 subjects; Test type: Superiority or Other; p < 0.001, Fisher Exact — A fixed sequence test procedure was used to control the study level type I error. Order of test sequence started with the primary efficacy endpoint and proceeded to the 3 secondary efficacy endpoints, in the order defined in the protocol; The 2-sided Fisher's Exact test was utilized to test for difference between NPSP558 and the placebo treatment groups; Treatment difference = 52.3, 95% CI 2-sided [40.6 to 64.0] — The above two sided asymptotic 95% confidence interval is based on normal approximation

2. Secondary Outcome: Percentage Changes From Baseline in Daily Calcium Dose at Week 24.
Description: The analysis of this endpoint was based on investigator prescribed data.
Time Frame: 24 Weeks
Population: Intent to Treat (ITT) population subjects with Baseline and Week 24 data
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Placebo | NPSP558
Number analyzed (Participants) | 33 | 79
percentage change from baseline | 2.4 (38.37) | -51.8 (45.71)
Statistical Analysis 1: Comparison: Placebo vs NPSP558; The null hypothesis is that there is no difference between the percentage changes from baseline for the two treatment arms; Test type: Superiority or Other; p < 0.001, ANCOVA — Following fixed sequence test procedure described in the primary endpoint section, statistical hypothesis testing was conducted for this secondary endpoint after the testing for the primary endpoint reached statistical significance; ANCOVA analysis conducted using percentage change from baseline as dependent variable, treatment as factor, and baseline calcium dose as covariate

3. Secondary Outcome: Proportion of Subjects Who Achieved Independence From Active Vitamin D and an Oral Calcium Dose of ≤ 500 mg/Day at Week 24.
Description: Subjects Who Achieved Independence from Active Vitamin D Usage and with Calcium Dose of 500 mg/day or less. This analysis was based on Investigator Prescribed Data.
Time Frame: 24 Weeks
Population: Intent to Treat (ITT) population subjects with Baseline and Week 24 data.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | NPSP558
Number analyzed (Participants) | 33 | 79
percentage of participants | 6.1 | 43.0
Statistical Analysis 1: Comparison: Placebo vs NPSP558; The null hypothesis is that there is no difference between the proportions of subjects (who achieved this secondary endpoint) from the two treatment arms; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Following fixed sequence test procedure described in the primary endpoint section, statistical hypothesis testing was conducted for this secondary endpoint after the testing for the first secondary endpoint reached statistical significance; Odds Ratio (OR) = 11.711, 95% CI 2-sided [2.619 to 52.363]

4. Secondary Outcome: Percentage of Subjects With Any Clinical Symptoms of Hypocalcemia During Weeks 16-24.
Description: Clinical symptoms were a selected group of adverse events that occurred during study weeks 16 through 24. The group of terms were defined by key opinion leaders and documented in study protocol.
Time Frame: 8 Weeks
Population: Intent to Treat (ITT) population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | NPSP558
Number analyzed (Participants) | 40 | 84
percentage of participants | 37.5 | 34.5
Statistical Analysis 1: Comparison: Placebo vs NPSP558; The null hypothesis is that the percentages of subjects with any reported clinical symptoms for the two treatment arms are the same; Test type: Superiority or Other; p = 0.747, Cochran-Mantel-Haenszel — Following fixed sequence test procedure described in the primary endpoint section, statistical hypothesis testing was conducted for this secondary endpoint after the testing for the second secondary endpoint reached statistical significance; Odds Ratio (OR) = 0.879, 95% CI 2-sided [0.402 to 1.922]

ADVERSE EVENTS:
Time Frame: 28 weeks
Description: 24 weeks on treatment plus 4 week follow-up period
Arm/Group | Placebo | NPSP558
Serious Adverse Events (participants affected / at risk) | 4/40 | 9/84
Other Adverse Events (participants affected / at risk) | 38/40 | 69/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=40) | NPSP558 (N=84)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Epididymal tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=40) | NPSP558 (N=84)
Paraesthesia (Nervous system disorders) | 10 (16) | 30 (69)
Hypocalcaemia (Metabolism and nutrition disorders) | 9 (10) | 33 (54)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12 (21) | 25 (41)
Nausea (Gastrointestinal disorders) | 7 (9) | 17 (35)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 8 (8)
Fatigue (General disorders) | 8 (11) | 10 (25)
Sinusitis (Infections and infestations) | 2 (2) | 6 (6)
Headache (Nervous system disorders) | 10 (20) | 22 (56)
Hypoaesthesia (Nervous system disorders) | 5 (6) | 16 (24)
Hypercalcaemia (Metabolism and nutrition disorders) | 4 (4) | 14 (17)
Tetany (Metabolism and nutrition disorders) | 4 (13) | 10 (24)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 10 (18)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 9 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 8 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (13)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 10 (13)
Vomiting (Gastrointestinal disorders) | 0 (0) | 10 (12)
Paraesthesia oral (Gastrointestinal disorders) | 3 (6) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 7 (9)
Hypercalciuria (Renal and urinary disorders) | 0 (0) | 6 (7)
Blood 25-hydroxycholecalciferol decreased (Investigations) | 0 (0) | 5 (5)
Anxiety (Psychiatric disorders) | 0 (0) | 5 (5)
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5)
Hypertension (Vascular disorders) | 2 (2) | 5 (5)
Dizziness (Nervous system disorders) | 3 (4) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Cystitis (Infections and infestations) | 2 (2) | 0 (0)
Herpes Zoster (Infections and infestations) | 2 (2) | 0 (0)
Viral Infection (Infections and infestations) | 2 (2) | 0 (0)
Injection Site Haematoma (General disorders) | 5 (6) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Feeling Cold (General disorders) | 2 (2) | 0 (0)
Oedema Peripheral (General disorders) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Urine Calcium Increased (Investigations) | 2 (3) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other